CLINICAL TRIAL: NCT00235950
Title: A Multicentre Study Comparing the Efficacy of Rosuvastatin With Atorvastatin When Given for a Period of 16 Wks to Subjects With Coronary Heart Disease & a Previously Performed Percutaneous Coronary Intervention
Brief Title: Assessment of the Lipid Lowering Effect of Rosuvastatin Compared to Atorvastatin in Subjects With Coronary Heart Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: D3560L00039
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Heart Disease; Percutaeous Coronary Intervention (PCI)
MeSH Terms: conditions — Coronary Disease | interventions — Rosuvastatin Calcium; Atorvastatin; Simvastatin; Clopidogrel

INTERVENTIONS:
Drug: Rosuvastatin or atorvastatin or simvastatin and clopidogrel
  Other Names: Crestor

SUMMARY:
The purpose of this study is to compare the efficacy between two lipid lowering treatments, rosuvastatin (10-40 mg) and atorvastatin (20-80 mg) in reducing low-density lipoprotein cholesterol (LDL-C) levels after 16 weeks of treatment in patients with coronary heart disease

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, established coronary heart disease with a previously performed PCI, previous treatment with clopidogrel, ongoing statin treatment, LDL-C>2.9 mmol/L, signed informed consent.

Exclusion Criteria:

* Ongoing treatment with clopidogrel for more than 12 weeks after randomisation, hypersensitivity to any of the study drugs, active liver disease, moderate or severe renal impairment, hereditary for or known muscular or neuromuscular disease and/or increased serum CK, pregnancy or lactation or of childbearing potential not practising an adequate method of contraception, use of concomitant medication with possible interaction with

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255
Dates: Start 2004-01; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of once daily treatment with rosuvastatin with the efficacy of treatment with atorvastatin

SECONDARY OUTCOMES:
Compare the impact of treatment with rosuvastatin to that of atorvastatin and simvastatin on clopidogrel initiated inhibition of platelet aggregation in a subset of subjects recruited in the Stockholm region.
Compare the impact of treatment with rosuvastatin to that of atorvastatin on clopidogrel initiated inhibition of platelet aggregation in all subjects, totally and on each dose of rosuvastatin and atorvastatin.
Compare the efficacy of treatment with rosuvastatin with the efficacy of treatment with atorvastatin in reducing LDL-C levels
Compare the efficacy of once daily treatment with rosuvastatin with that of atorvastatin in modifying levels of TC, HDL-C, TG, nonHDL-C (TC-HDL-C), LDL-C
Compare the titration schedule of rosuvastatin with that of atorvastatin.
Determine the safety by evaluating the incidence and severity of adverse events and abnormal laboratory values through 16 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Medical Science Director, MD, Study Director — AstraZeneca
Locations (18):
- Sweden (18):
  - Research Site, Danderyd
  - Research Site, Eksjö
  - Research Site, Falun
  - Research Site, Gothenburg
  - Research Site, Helsingborg
  - Research Site, Jönköping
  - Research Site, Karlskrona
  - Research Site, Karlstad
  - Research Site, Ljungby
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Örebro
  - Research Site, Skövde
  - Research Site, Stockholm
  - Research Site, Sundsvall
  - Research Site, Uppsala
  - Research Site, Vaxjo
  - Research Site, Västerås